CLINICAL TRIAL: NCT01340742
Title: Remote Ischemic Preconditioning Before Abdominal Surgery and the Prevalence of Perioperative Complications
Brief Title: Remote Ischemic Preconditioning Before Abdominal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R-10-132; 16811 (Other: REB)
Record Dates: First submitted 2011-02-14; First posted 2011-04-25 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Remote ischemic preconditioning; Abdominal surgery; Perioperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Arm remote preconditioning
  Interventions: Procedure: Remote Ischemic Pre-conditioning
- 2 (Placebo Comparator): Control group.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote Ischemic Pre-conditioning — Cuff placed on arm. Three 5- minute cycles of blood pressure cuff inflation: cuff is inflated to 200 mm Hg for 5 minutes followed by a 5-minute deflation (reperfusion.)
  Arms: 1
Procedure: Control — Cuff placed on arm uninflated for 30 minutes.
  Arms: 2

SUMMARY:
Major abdominal surgeries are associated with perioperative cardiac morbidity of up to 10%.

Ischemic preconditioning may have a protective effect. The purpose of this study is to find out remote ischemic conditioning by inflating a blood pressure cuff on the arm will have a protective effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery:large bowel, pancreatic and hepatic surgery

Exclusion Criteria:

* Chronic inflammatory disease.
* Glyburide use before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Events: incidence of MI, TIA/stroke, death in both groups | One week

SECONDARY OUTCOMES:
Renal function deterioration in the first week after surgery | One week
  Baseline Creatinine levels will be compared to the highest creatinine levels noted in the first 7 days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Lavi, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada